CLINICAL TRIAL: NCT06743932
Title: A Prospective Cohort Study of Combined Subinguinal Varicocele Ligation and Sclerotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mostafa Khedr, resident doctor at Assiut University hospital, Assiut University
Other Study IDs: VC Ligation + Sclerotherapy
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Varicocele
Keywords: Ligation; Sclerotherapy
MeSH Terms: conditions — Varicocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- varicocel patients: varicocele patients will be follow up after Ligation and Sclerotherapy

SUMMARY:
Traditional surgical ligation of the spermatic cord veins is effective in reducing the size of the varicocele and improving fertility outcomes. However, this procedure can be associated with complications such as hydrocele formation and recurrence . Antegrade sclerotherapy offers a minimally invasive alternative, involving the injection of a sclerosing agent directly into the dilated veins to achieve occlusion and reduce reflux .

This study aims to optimize treatment outcomes for varicocele by combining the benefits of surgical ligation with the sclerosing effects of sclerotherapy .The primary goal is to evaluate the efficacy and safety of combining antegrade sclerotherapy and surgical ligation in the treatment of varicocele .

DETAILED DESCRIPTION:
Varicocele (VC) is a vascular condition characterized by the abnormal development or blockage of veins in the scrotum, resulting in dilation, elongation, and twisting of the veins in the spermatic cord. Clinically, VC can cause scrotal pain, discomfort, and progressive testicular dysfunction. The prevalence of clinically diagnosed varicocele is approximately 8-16% in adolescents and 15% in adults. VC is a common and correctable cause of male infertility, responsible for around 44% of primary infertility cases . Other reports suggest that the prevalence in childhood and adolescence is similar to that in adulthood. A recent European study of 7,000 young men (median age: 19 years) reported a 15.7% prevalence of varicocele .

Severe and prolonged VC can lead to significant damage to the testes and accessory structures, causing 45-81% of secondary infertility cases. VC most commonly occurs on the left side (77-92% of cases) due to the anatomy of the left internal spermatic vein. Bilateral VC is observed in 10% of cases, while isolated right-sided VC is rare (1%). The diagnosis of VC is primarily based on physical examination, often supplemented by imaging . The American Society for Reproductive Medicine and the Society for Male Reproduction and Urology recommend treating VC favorably, even in the absence of severe symptoms, if it poses a risk for infertility or decreased semen quality. Treatment options for VC include general management (lifestyle modifications, physiotherapy), medication (for varicose symptoms, pain relief, and improvement in semen quality), and various surgical approaches (ligation of the internal spermatic vein via inguinal, retroperitoneal, or subinguinal routes) . Minimally invasive techniques, such as laparoscopy, surgical microscopy, and percutaneous embolization, have been developed to improve visualization and reduce surgical trauma.

ELIGIBILITY:
Inclusion Criteria:

* 1- Clinically and Doppler confirmed grades II or III varicocele. 2- All left, right or bilateral side varicocele. 3- Testicular pain or testicular atrophy. 4- Presence of at least one impaired semen parameter. 5- Age more than 18years

Exclusion Criteria:

* 1- Pre-existing hydrocele. 2- Concomitant hernia 3- Previous inguinal surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — male
Study Population: varicocele patients withClinically and Doppler confirmed grades II or III varicocele.
Sampling Method: Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
varicocele grade | 30 day
  Assess the change in varicocele grade from baseline to post-treatment using clinical examination and/or ultrasound

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abd Ellatif ME, Asker W, Abbas A, Negm A, Al-Katary M, El-Kaffas H, Moatamed A. Varicocelectomy to treat pain, and predictors of success: a prospective study. Curr Urol. 2012 May;6(1):33-6. doi: 10.1159/000338867. Epub 2012 Mar 18. PMID 24917707
- [Background] Su JS, Farber NJ, Vij SC. Pathophysiology and treatment options of varicocele: An overview. Andrologia. 2021 Feb;53(1):e13576. doi: 10.1111/and.13576. Epub 2020 Apr 9. PMID 32271477